CLINICAL TRIAL: NCT05655234
Title: Effect of Music Breathing, a Programme Based on Mindful Breathing and Music Therapy for Promoting Sense of Coherence in Young People: A Randomized Controlled Trial
Brief Title: Effect of Music Breathing for Promoting Sense of Coherence in Young People: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tung Wah College (Other)
Collaborators: Caritas Institute of Higher Education (Other)
Responsible Party: Principal Investigator, Winnie CHENG Lai Sheung, Professor of Practice, Caritas Institute of Higher Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UGC/FDS17(11)/H03/22
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Sense of Coherence
Keywords: music therapy; Sense of coherence; Mental well-being; Stress; Mindfulness; Randomized controlled trial
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We will conduct randomised controlled trial (RCT) to evaluate the effects of the MB programme
Who Masked: Outcomes Assessor
Masking Description: A research team member will be masked when performing data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving the MB programme (Experimental): Participants receiving the MB programme:
  meditative breathing; breathing while listening to music; drawing of a mental image while breathing; and processing and sharing of the experience. home practice
  Interventions: Behavioral: Music Breathing
- Participants receiving the control condition (Placebo Comparator): Mental health education programme:
  breathing exercise; stress reduction talk
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Music Breathing — The MB programme consists of four stages: 1. Silent breathing for grounding (SB), 2. Music breathing for grounding (MBG), 3. Music breathing for modulation (MM), 4. Music breathing for working (MW).
  After completing the silent breathing and music breathing practices, the participants will draw pictures of their body images of breathing space and centre. The form of the imagined breathing space expressed in the drawing and the meaning and content of the experience will be explored through a process facilitated by the therapist. The therapist's understanding of the participants' difficulties and progress will guide the next step, particularly the selection of music for the next sessions. The whole session takes about 2 hours. Weekly home practice is advised.
  Arms: Participants receiving the MB programme
Behavioral: Control condition — The control condition consists of 30-min mental health education programme with topics on stress management, music playing, and breathing exercise provided in the first and 6th weeks. A take-home kit which consists of the fact sheet information of the health talk and the video link of the breathing exercise and musical pieces will be provided to the participants after the first meeting. They are instructed to practice the breathing exercise and listening to the musical pieces at home.
  Arms: Participants receiving the control condition

SUMMARY:
The goal of this experimental study is to test the effects of Music Breathing (MB) in promoting a sense of coherence among young people.

The main questions it aims to answer are:

* What is the effect of a MB programme on personal resources (i.e., SOC, coping self-efficacy, emotion regulation and mindfulness) compared with the control condition in young people?
* What is the effect of a MB programme on stress reduction (i.e., depression, anxiety and stress, and salivary cortisol levels) compared with the control condition in young people? • • What is the effect of a MB programme on mental well-being compared with the control condition in young people?
* What is the relationship between SOC, coping self-efficacy, emotion regulation and mindfulness?

Participants will receive a MB programme in 6 weekly sessions and weekly home practice. The programme includes:

* meditative breathing;
* breathing with music listening;
* drawing a mental image of the breathing practice; and
* sharing and processing of the experience

DETAILED DESCRIPTION:
The proposed study will evaluate the effect of the Music Breathing (MB) programme on young people's sense of coherence in promoting coping with stress.

In the proposed randomised controlled trial, a sample of 290 young people (aged 18-30) will be recruited and allocated randomly into either the experimental or placebo control group. Participants in the experimental group will participate in a 6-week MB programme that will include music therapy and mindful breathing guided by a certified music therapist.

The following objectives are proposed:

* To examine the effect of a MB programme on promoting personal resources in young people;
* To examine the effect of a MB programme on reducing stress-related symptoms in young people; and
* To examine the effect of a MB programme on promoting mental well-being in young people.

This is a two-arm, parallel randomised controlled trial (RCT). Randomisation involving computer-generated two-digit random numbers (even and odd) (Excel 2007, Microsoft, Redmond, WA, USA) will be used to allocate participants in sequence to either the intervention group or control group in a 1:1 ratio after they have provided consent to participate. The allocation will be blinded to the participants and the data analyst. The random allocation will be conducted by a research assistant who will not be involved in the intervention and data analysis. Participants in the experimental arm will receive a 6-week MB programme. Participants in the control arm will placebo control programme and will be blinded to the study details. Data will be collected from both groups at three time points: before-intervention (T0), after-intervention (week 6; T1) and 1-month follow-up (week 10; T2), except the salivary cortisol levels which will be assessed at T0 and T1.

The participants will be recruited from universities and district centres through emails, social media, leaflets and posters. The estimated sample size has been calculated using the statistical package G*Power 3.1.9.4 (version 2019) for a multivariate analysis of variance (MANOVA) according to the effect size (Cohen's d) (between 0.43 and 0.59) of anxiety in previous study on group music-guided imagery (Torres et al., 2018). When converting to a repeated measure (Cohen's f), the effect size is considered moderate (f = 0.25), with a type I error rate of 5% (2-sided) and assuming a correlation of 0.5 between repeated measures. To achieve 90% power to measure outcome three times in two groups, 232 subjects (n=116 per group) will be required (Cohen, 1988). Assuming a 20% attrition rate (Porter et al., 2012), the trial will require at least 145 participants starting in each arm.

To ensure treatment fidelity, the certified music therapist will have at least 25 hours of MB programme training; the implementation of the intervention will be supervised by Dag Körlin, the Co-I. The group sessions will be audio-taped with the consent of the participants, and the recordings will be given to the supervisor for quality monitoring. Written session reports will be provided and regular meetings via Zoom (i.e., three supervisions in the first group, and then two supervisions in the subsequent groups) will be arranged for maintaining the quality of the intervention. The research team will discuss any issues that may arise regarding the study protocol to ensure the quality and consistency of study intervention via regular face-to-face or online meetings.

Ethical clearance has been obtained prior to the study from the study institution. Consent will be obtained and anonymity ensured to protect privacy. Participants will receive study information and have autonomy to withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* moderate stress level measured with perceived stress scale (PSS-10) >or =14-26
* a liking for music

Exclusion Criteria:

* diagnosed with an acute mental problem;
* participants under the influence of drugs that affect the nervous system;
* having previous experience with imagery evoked by music and meditations where music is played.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sense of coherence: change from pre-intervention to post-intervention in sense of coherence | Pre- to post-intervention (10 weeks)
  The 13-item Chinese version of the Sense of Coherence Scale (C-SOC-13) ranges from 1 to 7. Higher scores indicate greater levels of sense of coherence.

SECONDARY OUTCOMES:
Coping self-efficacy: change from pre-intervention to post-intervention in coping self-efficacy | Pre- to post-intervention (10 weeks)
  The 26-item Coping Self-Efficacy Scale (CSES) ranges from 0-10. Higher scores indicate greater levels of coping self-efficacy.
Emotion regulation: change from pre-intervention to post-intervention in emotion regulation | Pre- to post-intervention (10 weeks)
  The 36-item Difficulties in Emotion Regulation Scale (DERS) ranges from 1 to 5. Higher scores indicate more difficulty in emotion regulation.
Mindfulness: change from pre-intervention to post-intervention in mindfulness | Pre- to post-intervention (10 weeks)
  The 15-item Mindful Attention Awareness Scale (MAAS) (Chinese version) ranges from 1-6. Higher scores reflect higher levels of dispositional mindfulness.
Depression, anxiety and stress: change from pre-intervention to post-intervention in depression, anxiety and stress | Pre- to post-intervention (10 weeks)
  The 21-item Depression Anxiety Stress Scales (DASS-21) (Chinese version) range from 0-3.
  Higher scores reflect higher levels of depression, anxiety, and stress.
Subjective general well-being; change from pre-intervention to post-intervention in subjective general well-being | Pre- to post-intervention (10 weeks)
  The 24-item BBC Subjective Well-being Scale (BBC-SWB) ranges from 1-5. The higher score indicates better levels of well-being.
Salivary cortisol | post-intervention at week 6
  Salivary cortisol levels (sCort)

OTHER OUTCOMES:
Demographic information | before the intervention
  A self-developed questionnaire will be used to collect demographic information about the participants, including age, gender, educational level, religious beliefs and practices, socioeconomic status and coping behaviour. The latter will be assessed using the Brief Cope Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Winnie LS Cheng, PhD, Principal Investigator — Caritas Institute of Higher Education

IPD SHARING:
Plan to Share IPD: No
The data can be released when requested.

REFERENCES:
- [Derived] Cheng WL, Tang AC, Tsang MC, Wong LL, Korlin D. Effect of music breathing, a program based on mindful breathing and music listening therapy for promoting sense of coherence in young people: study protocol for a randomized controlled trial. Trials. 2023 Oct 12;24(1):662. doi: 10.1186/s13063-023-07645-x. PMID 37828487

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT05655234/Prot_SAP_000.pdf